CLINICAL TRIAL: NCT05450276
Title: Patient-Reported Outcome Study of Project ECHO for ILD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Pulmonary Care and Research Collaborative Limited (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ILDC-003
Record Dates: First submitted 2022-06-30; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Interstitial Lung Disease
Keywords: Progressive Fibrosing Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease Associated With Systemic Sclerosis; Myositis-Associated Interstitial Lung Disease; Sarcoidosis; Hypersensitivity Pneumonitis; Pulmonary Fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Sarcoidosis; Alveolitis, Extrinsic Allergic; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will assess whether patients of providers participating in Project ECHO for ILD experience reduced stress, including financial stress, based on their ability to receive timely and local care and services, The study will employ nested mixed-method design at baseline, at 6 months and at 12 months to answer the study question.

DETAILED DESCRIPTION:
Project ECHO (Extension for Community Healthcare Outcomes) is a knowledge-sharing model to expand the capacity of the health care workforce so that more people can get high quality care for their health conditions in or near the communities where they live. The model brings specialty disease expertise to community providers through its hub-and-spoke networks. The model relies on videoconferencing to connect local providers in non-urban or underserved communities (spoke sites) with an interdisciplinary team of specialist providers at academic medical centers (hubs) during virtual "teleECHO" clinic sessions, which include brief educational lectures and case-based, experiential learning.

The ECHO model addresses barriers of long wait times for a first appointment, the time and expense associated with long distance travel, and the disinclination to follow through on repeated care appointments in the face of these persistent barriers, all with the additional objective of achieving health equity. Most patients perceive the diagnostic and care pathways in ILDs as a major struggle because of lack of awareness about the diseases, delayed access to specialty centers, providers' focus on disease- versus patient-centered care, and lack of reliable information and education about the diseases and supportive care resources.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of interstitial lung disease
* Not be currently followed by an ILD specialist at an academic institution or must live more than 50 miles away from an academic ILD center

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of pulmonologists and primary care physicians who participate in Project ECHO for ILD.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in patients' stress level | Up to 18 months
  Assessed by the Perceived Stress Scale at baseline, 6 months, and at study end. The range of scores is 0-40, with higher scores indicating more appraised stress.
Patients' satisfaction of care | Up to 18 months
  Assessed by the Patient Satisfaction Survey, a self-report scale assessing patient experience and satisfaction with local ILD care, which is composed of 28 items rated on a Likert Scale and Yes/No grading; the summed items produce a single satisfaction score.

SECONDARY OUTCOMES:
Change in patients' perceptions regarding local ILD care | Up to 18 months
  Patient participants in the study will complete interviews at baseline (their community PCP or pulmonologist attending their first ILD teleECHO clinic), at 6 months and at 12 months. The interviews will be open-ended to solicit the perspectives of participants regarding their experience with the local ILD care in their communities before, during and after their PCPs or local pulmonologists participate in Project ECHO for ILD.

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Barakat, PhD, Principal Investigator — Pulmonary Care and Research Collaborative, Ltd.
Locations (1):
- Pulmonary Care and Research Collaborative, Ltd., Boston, Massachusetts, United States